CLINICAL TRIAL: NCT00314340
Title: A CTSC Clinical Research Center Study: A Comparison of the Addiction Liability of Hydrocodone and Sustained Release Morphine
Brief Title: A Comparison of the Addiction Liability of Hydrocodone and Sustained Release Morphine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 200513430
Record Dates: First submitted 2006-04-11; First posted 2006-04-13 (Estimated); Results first posted 2013-07-12 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Chronic Pain
Keywords: Chronic Pain; Opioids
MeSH Terms: conditions — Chronic Pain | interventions — Ethanol; benzedrine; Amphetamine; Hydrocodone; Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- extended-release morphine (Active Comparator): Markers of Abuse Liability, Neuropsych Testing, and Cue Reactivity
  On one of three study dates, subjects received ER morphine tablets, 45 mg (Mallinckrodt Pharmaceuticals, St. Louis, MO). The dose of ER morphine sulfate (45 mg) was selected because of its approximate equianalgesic effect to the dose of hydrocodone-acetaminophen (30/925 mg).
  Interventions: Behavioral: Markers of Abuse Liability, Neuropsych Testing, and Cue Reactivity; Drug: ER Morphine
- hydrocodone (Active Comparator): Markers of Abuse Liability, Neuropsych Testing, and Cue Reactivity
  On the day of the study session, patients received hydrocodone 30 mg plus N-acetyl-para-aminophenol 975 mg (APAP;Qualitest Pharmaceuticals Inc, Huntsville, AL).
  Interventions: Behavioral: Markers of Abuse Liability, Neuropsych Testing, and Cue Reactivity; Drug: hydrocodone plus acetaminophen
- placebo (Placebo Comparator): Subjects received a placebo pill if randomized to this arm. Both opioid medications and the placebo were administered in identical capsules.
  Interventions: Behavioral: Markers of Abuse Liability, Neuropsych Testing, and Cue Reactivity; Drug: placebo

INTERVENTIONS:
Behavioral: Markers of Abuse Liability, Neuropsych Testing, and Cue Reactivity — The first dose of the study medication was taken following collection of baseline measurements, and subsequent measurements were taken hourly thereafter. Respiration, heart rate, arterial oxygen saturation (pulse oximetry), and blood pressure were also monitored at these intervals to insure the safety of subjects.
  Other Names: Craving for drugs on 5 visual analog scales; Addiction Research Center; Morphine-Benzedrine Group (euphoria); Phenobarbital-Chorpromazine-Alcohol (sedation); Lysergic Acid Diethylmide (dysphoria, agitation); Benzedrine (an empiric amphetamine scale); Amphetamine (activation); Cue reactivity testing; Neurocognitive testing
Drug: ER Morphine
  Other Names: extended release morphine
  Arms: extended-release morphine
Drug: hydrocodone plus acetaminophen
  Arms: hydrocodone
Drug: placebo
  Arms: placebo

SUMMARY:
Characterize the relative abuse liability of a short versus a long acting opioid in chronic pain patients.

DETAILED DESCRIPTION:
A placebo-controlled, double-blind, crossover trial will be conducted providing study subjects either hydrocodone/acetaminophen 30mg/975mg, sustained release morphine 45mg or placebo on separate GCRC visits. A long acting comparator (slow-release morphine sulfate 45 mg) will be chosen because of its putative equianalgesic effects to the dose of hydrocodone (30 mg) selected. Subjects will participate in the three sessions at the UC Davis/Mather Medical Center General Clinical Research Center (GCRC) at intervals of 7-10 days. Sessions will be approximately 360 min in duration. Subjects will receive either hydrocodone/acetaminophen or sustained release morphine around-the-clock for 7-10 days prior to the experimental session. At each experimental session, an assessment of abuse liability will be completed before the intake of medications, as well as at 0, 60, 120, 180, 240 minutes after the ingestion of the study medication.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic pain for periods greater than 6 months
* Patients taking greater than 80 mg morphine equivalents of a short acting opioid (>8 vicodin or 4 oxycodone/day)
* Referral to Pain or Substance Abuse Clinic for self-escalation of opioids

Exclusion Criteria:

* Inability to understand and comprehend spoken English
* Patients with Munchausen's syndrome
* Patient has a history of Peripheral Vascular Disease
* Patient has a history of Raynaud's Phenomenon
* Liver Disease; Child's classification greater than 1 (liver cirrhosis) will be excluded
* Renal disease (BUN >25 or Cr >1.5)
* Congestive Heart Failure; Subjects with New York Heart Association (NYHA)Heart Failure Symptom Classification System Level of Impairment II, III and IV will be excluded
* Coronary artery disease; recent MI within the past six months or recent history of angina not controlled with NTG within the past six months
* Hypertension; 1)previously normotensive subject; systolic bp >140 mm Hg and diastolic bp > 90 mm Hg 2) Hx of active treatment with antihypertensive medications; systolic bp >150 mm Hg and diastolic bp > 100 mm Hg
* Cerebrovascular disease; recent history within the past year of a transient ischemic attack or recent history within the past year of a cerebrovascular event
* Malignancy requiring active treatment
* Patient is pregnant (as ascertained by a self-report and a mandatory commercial pregnancy test before any study medication is consumed)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2005-11; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barth L Wilsey, MD, Principal Investigator — University of California, CA Medical Center Division of Pain Medicine

REFERENCES:
- [Result] Wilsey BL, Fishman S, Li CS, Storment J, Albanese A. Markers of abuse liability of short- vs long-acting opioids in chronic pain patients: a randomized cross-over trial. Pharmacol Biochem Behav. 2009 Nov;94(1):98-107. doi: 10.1016/j.pbb.2009.07.014. Epub 2009 Aug 4. PMID 19660492

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from the UC Davis Medical Center Pain and VA Northern California Pain Clinics in 2007-8. They had to have had chronic pain for more than 3 months and to have self-escalated their dose of a short-acting opioid (i.e., a combination product containing hydrocodone, codeine, or oxycodone)prescribed to treat their pain.
Pre-assignment Details: Of 55 patients approached, 18 were evaluated, and 14 met entry criteria and were enrolled. Two withdrew before starting the study. One subject withdrew after starting the study because of insufficient pain relief from the study medications leaving 35 visits by 12 patients for analysis.
Groups:
- All Participants: All participants were randomized to receive the ER morphine tablets, 45 mg, hydrocodone 30 mg plus N-acetyl-para-aminophenol 975 mg, or placebo in a 3 way cross over design.
Period: Overall Study
Arm/Group | All Participants
Started | 12
ER Morphine | 11
Hydrocodone Plus APAP | 12
Placebo | 12
Completed | 11
Not Completed | 1
Not completed — lost interest | 1

BASELINE CHARACTERISTICS:
Groups:
- Prescription Opioid Abusers: The subjective effects of the study drug were evaluated with the short form of the Addiction Research Center Inventory (ARCI. This inventory consists of 49 true/ false questions which survey major domains of drug effects. Participants indicated the pleasurable effects or desirability of the medications on 4 locally developed drug-liking ratings: craving, liking, strong desire, and "want more pain medication." Ratings were made on a 100-mm VAS anchored with 0 at the low end and 10 at the high end. Participants also responded to 11 locally developed drug-effect ratings to assess psychoactive effects. Ratings were again made on a 100-mmVAS anchoredwith 0 at the lowend and 10 at the high end for:"on cloud 9," "high," "good drug effect," "bad drug effect," "impaired,""stoned," "sedated," "confused," "nauseated from," "anxious," and "down". The rating levels over a six hour period were examined to explore the timing of these effects.
Arm/Group | Prescription Opioid Abusers
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 46 (4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 8
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: 3 Scores on the Addiction Research Center Inventory (ARCI)
Description: The subjective effects of the study drug were evaluated with 3 subscales of the Addiction Research Center Inventory (ARCI). The subscales studied included Morphine-Benzedrine Group which measured euphoria (0-16 with higher numbers indicating more euphoria), the Phenobarbital-Chorpromazine-Alcohol Group which measured sedation (-3 to +11 with higher scores indicating more sedation), and the Lysergic Acid Diethylmide Group which measured dysphoria and agitation (-4 to +10 with higher scores indicating more dysphoria). This inventory consists of 49 true/ false questions which survey major domains of drug effects. The ARCI was measured at six timepoints. Of interest were trough sedation, peak euphoria, and trough dysphoria.
Time Frame: 0, 60, 120, 180, 240, or 300 minutes
Population: Treatment effects at baseline, 60, 120, 180, 240, and 300 min were assessed with repeated measures ANOVA. A liner mixed-effects model with inclusion of interaction terms (1) treatment and time and (2) random order visit number and time was performed.
Measure: Mean (Standard Deviation); unit: scores on a scale
Groups:
- ER Morphine Tablets, 45mg: Scores of the 5 Addiction Research Center Inventory dimensions did not change significantly between baseline and 300 min under any treatment condition.
- Hydrocodone 30 mg Plus N-acetyl-para-aminophenol 975 mg: These findings all argue against the hypothesis that the hydrocodone product induced a greater euphoric or reinforcing effect than that of ER morphine.
Arm/Group | ER Morphine Tablets, 45mg | Hydrocodone 30 mg Plus N-acetyl-para-aminophenol 975 mg | Placebo
Number analyzed (Participants) | 11 | 12 | 12
scores on a scale
  trough sedation | 7.6 (1) | 5.4 (0.9) | 5.2 (0.8)
  peak euphoria | 3.3 (0.8) | 4.6 (0.9) | 3.5 (1.0)
  trough agitation | 4.7 (0.8) | 4.2 (0.6) | 3.6 (0.5)

ADVERSE EVENTS:
Arm/Group | Prescription Opioid Abusers
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No